CLINICAL TRIAL: NCT06562608
Title: Neural Mechanisms of Anticholinergic Burden in Mid- to Late-Life Schizophrenia Spectrum
Brief Title: Anticholinergic Deprescription in Schizophrenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Deepak K. Sarpal, M.D. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Deepak K. Sarpal, M.D., Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY24050090; R01MH135096 (NIH)
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Anticholinergic Deprescription (Experimental): In this arm, clinically determined unneeded benztropine or trihexyphenidyl will be deprescribed, per routine care by clinical providers.
  Interventions: Drug: Anticholinergic Deprescription
- No Anticholinergic Deprescription (Active Comparator): In this arm, no deprescription of benztropine or trihexyphenidyl will occur.
  Interventions: Drug: No Anticholinergic Deprescription
- Healthy Controls (No Intervention): In this arm, a healthy control group with minimal anticholinergic burden will be examined longitudinally.

INTERVENTIONS:
Drug: Anticholinergic Deprescription — per routine clinical care, people in the active arm of the study will undergo deprescription of benztropine or trihexyphenidyl per routine clinical care.
  Arms: Anticholinergic Deprescription
Drug: No Anticholinergic Deprescription — In this arm, no deprescription of benztropine or trihexyphenidyl will occur.
  Arms: No Anticholinergic Deprescription

SUMMARY:
In this study, the investigators will examine whether a deprescription of unnecessary anticholinergic drugs (benztropine or trihexyphenidyl) can augment quality of life, functioning, and neurocognition in individuals who with schizophrenia. Individuals identified by clinical services who have unneeded prescriptions benztropine or trihexyphenidyl will be eligible for deprescription and study entry. Following a baseline evaluation and magnetic resonance imaging (MRI), participants will will be randomized to either staying on their anticholinergic drugs or undergoing deprescription per routine clinical care, and will undergo follow-up evaluations across 6 months. The investigators predict that reducing and deprescribing these drug, if clinically determined to be unnecessary will will enhance functioning, neurocognition

ELIGIBILITY:
Inclusion Criteria:

1. Primary DSM-defined diagnosis of schizophrenia or schizoaffective disorder verified by the Structured Clinical Interview for DSM-5 (SCID).
2. Prescription of benztropine or trihexyphenidyl for at least 6 months
3. Age 40-70 years.
4. ACBS score >= 3.
5. Mild or absent extrapyramidal symptoms (Determined by clinical pharmacists and prescribers).
6. Competency and willingness to sign informed consent.

Inclusion criteria for the healthy control group:

1. Age 40-70 years.
2. Competency and willingness to sign informed consent.

Exclusion Criteria:

1. Serious anticholinergic side-effects (e.g., fever, blurred vision) indicative of a need for immediate removal of anticholinergics,
2. Serious neurologic or medical condition/treatment that impacts the brain and Neurodegenerative conditions such as Parkinson's, dementia, etc.; autoimmune conditions such as Multiple Sclerosis (MS) and lupus; as well as traumatic brain injury (TBI).
3. Significant risk of suicidal or homicidal behavior.
4. Cognitive or language limitations, or any other factor that would preclude subjects providing informed consent.
5. Contraindications for MR imaging (e.g., a pacemaker).
6. Current SCID-verified substance use disorder will be excluded to avoid the confounding impact of significant substance use comorbidity. Participants with a history of substance use disorder that is in early or full remission will be eligible, to enhance generalizability.
7. Patients concurrently treated with electroconvulsive therapy will be excluded because of its effects on cognition.

Exclusion criteria for Healthy Control (HC) subjects:

1. No history of psychotic illness and no active Axis I disorder as determined by clinical interview using the SCID-NP.
2. Score greater than 1 on the ACB scale.
3. MR imaging contraindications.
4. Neurologic conditions, any serious non-psychiatric disorder that could affect brain functioning, or intellectual disability.
5. HC with family history of psychosis will be excluded, as such individuals show subtle, but significant cognitive and neurobiological abnormalities.
6. Individuals currently taking anticholinergic medications for reasons other than SSD.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in cognitive performance via scores from the MATRICS Consensus Cognitive Battery.
Change in scores on quality of life assessments. | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in quality of life, measured with the WHOQOL-BREF.
Change in scores on functional outcome assessments. | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in functional outcomes, measured with the Specific Level of Functioning Scale.
change in brain functional connectivity. | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in brain functional connectivity between the basal forebrain and linked structures, such as regions of the cognitive control network, and the globus pallidus.
change in activation of neurocognitive networks | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in brain activation of the cognitive control network via the AX-CPT, and activation of the hippocampus during memory encoding/retrieval via the Relational and Item-Specific Encoding task.
Brain glutamate concentration | 6 months
  We will examine whether the anticholinergic deprescription group, relative to the non-deprescription group, shows an increase in brain glutamate concentrations in the hippocampus and the dorsal anterior cingulate cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Sarpal, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Western Psychiatric Hospital/University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data to the National Institute of Mental Health (NIMH) data archive
Supporting Information: Study Protocol, CSR, Analytic Code